CLINICAL TRIAL: NCT01219829
Title: Refining the Molecular Progression From Intraductal to Invasive Pancreatic Cancer: Correlating Genetic Profiles and Clinicopathological Phenotypes in Sporadic and Familial Pancreatic Adenocarcinoma
Brief Title: Pancreatic Intraepithelial Neoplasia (PanIN) and the Association With Recurrence of Pancreatic Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Cold Spring Harbor Laboratory (Other)
Responsible Party: Sponsor
Other Study IDs: AAAD5381
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic intraepithelial neoplasia (PanIN); Pancreatic Cancer; Recurrence of pancreatic cancer; Field Effect; Genetic mutations in pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — * Blood samples
  * Specimens of tumors, pre-cancerous lesions, and normal tissue from patients who need to have endoscopy or surgery for diagnosis or treatment of tumors that develop
  * Samples of urine and stool, and duodenal aspirates if an individual will be having an endoscopy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family History patients: Patients with a strong family history of pancreatic cancer or with a genetic syndrome that puts them at risk for pancreas cancer.
- Recurrence patients: Patients who underwent surgery for pancreatic cancer and developed tumor recurrence after surgery

SUMMARY:
The research purpose of this project is to create a registry, and blood and tissue bank for individuals at high-risk for pancreatic cancer. We plan to conduct histopathological and molecular analysis of resected pancreatic tissue prospectively collected from a cohort of pancreatic cancer patients.

DETAILED DESCRIPTION:
Pancreatic cancer is the fifth leading cause of cancer-related death in the United States. In order to improve outcomes of this disease, significant research efforts have focused on understanding the changes that occur in the pancreas prior to tumor occurrence. The types of changes most often associated with tumor have been named pancreatic intraepithelial neoplasia (PanIN). It is not yet clear how to identify the PanIN lesions most likely to develop into cancer and the length of time required for this progression. In order to evaluate these questions, we are interested in examining the microscopic and genetic characteristics of PanIN lesions in two "high-risk" patients: 1) patients who underwent surgery for pancreatic cancer and developed tumor recurrence after surgery and 2) patients with a strong family history of pancreatic cancer or with a genetic syndrome that puts them at risk for pancreas cancer. The surgical specimens from these patients will be evaluated by a pathologist for evidence of widespread PanIN lesions. In addition, PanIN lesions will be tested for abnormalities in several major genes that are known to be important in pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Tissue-confirmed diagnosis of pancreatic adenocarcinoma.
* Underwent surgical resection for adenocarcinoma at Columbia-Presbyterian Medical Center with pathologically negative surgical margins.
* Enrolled in our Pancreatic Cancer Registry and Tissue Bank protocol (AAAA-6154).
* Have at least 2 relatives (of whom one must be first-degree relative) with pancreatic cancer, or have been diagnosed with a a genetic syndrome which is associated with pancreatic cancer (among the included syndromes include BRCA1/2, FAMMM, Peutz-Jeghers, HNPCC, Hereditary Pancreatitis) -OR- Have radiological or pathological (fine needle aspirate or surgical biopsy) evidence of local tumor recurrence following surgery.

Exclusion Criteria:

* Metastatic disease discovered at presentation or on recurrence (exception is the familial PDC patients)
* Positive surgical margins.
* Lack of clinical followup at one year following surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are identified by a clinician as having either 1) a strong family history of pancreatic cancer; or 2) evidence (radiological or pathological) of local tumor recurrence following surgical resection, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2009-03-18 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Number of subjects with histological features of PanIN lesions assessed | 1 year
  Distinctive histological features of PanIN within surgical specimens of our two study groups will be assessed by pathologists.

SECONDARY OUTCOMES:
Evaluation of clonality multifocal PanIN lesions | 1 year
  Using microarray-based comparative genomic hybridization (aCGH) to evaluate the samples.
Evaluation of Recurrence Mechanism in PDC | 1 year
  aCGH will also be utilized to evaluate recurrence mechanism in a set of cases in which both original tumor and recurrence tumor was resected, allowing for clonal origins to be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy K Chung, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No